CLINICAL TRIAL: NCT02534480
Title: A Randomized, Placebo-Controlled, Double-Blind, Single Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Orally-administered NGP 555 in Healthy Young Volunteers
Brief Title: Neurogenetic Pharmaceuticals (NGP) 555 in Healthy Young Volunteers (Single-ascending Dose)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NeuroGenetic Pharmaceuticals Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NGP 555-001
Record Dates: First submitted 2015-04-27; First posted 2015-08-27 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Alzheimer's Disease
Keywords: Amyloid
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- NGP 555 25 mg (Active Comparator): NGP 555 25 mg capsule and placebo by mouth once per day
  Interventions: Drug: NGP 555
- NGP 555 50 mg (Active Comparator): NGP 555 50 mg capsule and placebo by mouth once per day
  Interventions: Drug: NGP 555
- NGP 555 100 mg (Active Comparator): NGP 555 100 mg capsule and placebo by mouth once per day
  Interventions: Drug: NGP 555
- NGP 555 200 mg (Active Comparator): NGP 555 200 mg capsule and placebo by mouth once per day
  Interventions: Drug: NGP 555
- NGP 555 300 mg (Active Comparator): NGP 555 300 mg capsule and placebo by mouth once per day
  Interventions: Drug: NGP 555

INTERVENTIONS:
Drug: NGP 555 — Gamma-secretase modulator for the treatment of Alzheimer's disease
  Other Names: NGP555

SUMMARY:
NGP 555 is a small molecule preventative therapy aimed at reducing Alzheimer's disease amyloid buildup by targeting Abeta 42 production.

DETAILED DESCRIPTION:
NGP 555 is a gamma-secretase modulator with a selective mechanism to reduce Abeta 42 while raising shorter Abeta forms such as Abeta 37 and 38.

NGP 555 is being developed as a preventative disease modifying therapy for Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female volunteers aged 18-55 yrs and in good health as determined by medical history, physical examination, clinical laboratory studies, electrocardiograms (ECGs), vital signs, and investigator judgment
2. Volunteer voluntarily agrees to participate in this study and signs an Institutional Review Board (IRB)-approved informed consent prior to performing any of the screening procedures
3. Female volunteers who are of child-bearing potential must agree to use a medically acceptable method of contraception (e.g., abstinence, an intrauterine device.
4. Male healthy volunteers willing to use barrier contraception.
5. Body mass index (BMI) of ≥ 18.0 kg/m2 and ≤ 32.0 kg/m2

Exclusion Criteria:

1. History of seizure disorder, symptomatic seizures (not including a history of simple febrile seizures in childhood) or any past or present medical condition which, in the opinion of the investigator has the potential to reduce seizure threshold (e.g., history of head trauma or concussion, previous alcohol abuse, substance abuse)
2. Any concurrent disease or condition that, in the opinion of the Investigator, would make the volunteer unsuitable for participation in the clinical study
3. History of alcohol and/or illicit drug abuse within two years of entry
4. Any psychiatric diagnosis or symptoms (e.g., hallucinations, major depression, anxiety or delusions)
5. History of cerebrovascular events or non-vasovagal related loss of consciousness
6. History of cardiac arrhythmias, ischemic heart disease or cerebrovascular disease
7. Hepatic impairment as defined by >1.3 times the upper limit of normal ranges of serum liver enzymes
8. Renal impairment as defined by abnormal ranges of serum creatinine.
9. Presence of clinically significant orthostatic hypotension (fall in systolic blood pressure of >20 mmHg or fall diastolic blood pressure of > 10 mmHg; and increase in heart rate by > 20 beats per minute [bpm])
10. Corrected QT interval (QTc) values of > 450 ms for males and > 470 ms for females.
11. Volunteers with abnormally low serum B12, folate or abnormal thyroid function tests
12. Positive Screening test for Hepatitis B surface antigen (HBsAg), Hepatitis C antibody, or human immunodeficiency virus (HIV) antibody
13. Positive urine test for alcohol or drugs
14. Suicidal ideation
15. Female volunteers that are breastfeeding or female volunteers with a positive urine pregnancy test
16. Clinically significant deviation from normal in physical examination, vital signs or clinical laboratory tests
17. Volunteer is unable to understand the protocol requirements, instructions and study-related restrictions, the nature, scope and possible consequences of the clinical study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-03; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events as a measure of safety and tolerability | 0-96 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Apinya Vutikullird, DO, Principal Investigator — WCCT
Locations (1):
- WCCT, Cypress, California, United States